CLINICAL TRIAL: NCT00070525
Title: A Phase II Study of R115777 (Zarnestra) (NSC # 702818, IND# 58,359) in Children With Recurrent or Progressive: High Grade Glioma, Medulloblastoma/PNET or Brainstem Glioma
Brief Title: Tipifarnib in Treating Young Patients With Recurrent or Progressive High-Grade Glioma, Medulloblastoma, Primitive Neuroectodermal Tumor, or Brain Stem Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01806; NCI-2012-01806 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000334862; COG-ACNS0226; ACNS0226 (Other: Children's Oncology Group); ACNS0226 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Childhood High-grade Cerebral Astrocytoma; Childhood Oligodendroglioma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Medulloblastoma; Optic Nerve Glioma | interventions — tipifarnib

ARMS (1):
- Arm I (Experimental): Patients receive oral tipifarnib twice daily on days 1-21. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib

INTERVENTIONS:
Drug: tipifarnib — Given orally

SUMMARY:
This phase II trial is studying how well tipifarnib works in treating young patients with recurrent or progressive high-grade glioma, medulloblastoma, primitive neuroectodermal tumor, or brain stem glioma. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate in pediatric patients with recurrent or progressive high-grade glioma, medulloblastoma/primitive neuroectodermal tumor (PNET), or brain stem glioma treated with tipifarnib.

II. Determine the distribution of time to progression, time to treatment failure, and time to death in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to disease (high-grade glioma vs recurrent or progressive medulloblastoma/primitive neuroectodermal tumor [PNET] vs progressive diffuse, intrinsic brain stem glioma).

Patients receive oral tipifarnib twice daily on days 1-21. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed brain tumor, including the following:

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic oligodendroglioma
  * Medulloblastoma/primitive neuroectodermal tumor (PNET)
  * Diffuse intrinsic brain stem glioma*
* Progressive or relapsed disease after prior conventional therapy
* Radiographic evidence of measurable disease
* Performance status - Karnofsky 60-100% (over 16 years of age)
* Performance status - Lansky 60-100% (16 years of age and under)
* Performance status - ECOG 0-2
* At least 8 weeks
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 8.0 g/dL (red blood cell transfusions allowed)
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGPT and SGOT less than 2.5 times ULN
* Creatinine clearance OR radioisotope glomerular filtration rate at least 70 mL/min
* Maximum creatinine based on age as follows:

  * 0.8 mg/dL (5 years and under)
  * 1.0 mg/dL (6 to 10 years)
  * 1.2 mg/dL (11 to 15 years)
  * 1.5 mg/dL (over 15 years)
* Shortening fraction at least 27% by echocardiogram
* Ejection fraction at least 50% by MUGA
* No dyspnea at rest
* No exercise intolerance
* Pulse oximetry greater than 94%*
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Seizure disorder is allowed provided it is well-controlled on non-enzyme-inducing anticonvulsants
* No active graft-versus-host disease
* No uncontrolled infection
* No allergy to azoles (e.g., ketoconazole, itraconazole, or fluconazole)
* Recovered from prior immunotherapy
* At least 7 days since prior antineoplastic biologic agents
* At least 1 month since prior autologous stem cell transplantation (SCT)
* At least 6 months since prior allogeneic SCT
* More than 1 week since prior growth factors
* No concurrent immunomodulating agents
* More than 2 weeks since prior myelosuppressive chemotherapy (4-6 weeks for nitrosoureas or temozolomide) and recovered
* No concurrent anticancer chemotherapy
* Concurrent dexamethasone allowed provided patient is on a stable or decreasing dose for at least 1 week prior to study entry
* Concurrent corticosteroids allowed only for treatment of increased intracranial pressure
* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 3 months since prior craniospinal radiotherapy
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* No concurrent palliative radiotherapy
* No prior initiation of therapy on another phase II study
* No concurrent participation in another therapeutic COG study
* No concurrent enzyme-inducing anticonvulsants
* No other concurrent anticancer or experimental drugs
* No concurrent foods or medications that interfere with CYP3A4, including any of the following:

  * Carbamazepine
  * Phenytoin
  * Phenobarbital
  * Grapefruit juice
  * Erythromycin
  * Azithromycin
  * Clarithromycin
  * Rifampin and its analogues
  * Fluconazole
  * Ketoconazole
  * Itraconazole
  * Cimetidine
  * Cannabinoids (i.e., marijuana or dronabinol)
  * Omeprazole
  * Hypericum perforatum (St. John's wort)
  * Ethosuximide
  * Glucocorticoids
  * Griseofulvin
  * Nafcillin
  * Nelfinavir
  * Norfloxacin
  * Norfluoxetine
  * Nevirapine
  * Oxcarbazepine
  * Phenylbutazone
  * Primidone
  * Progesterone (all progestins)
  * Rifabutin
  * Rofecoxib
  * Sulfadimidine
  * Sulfinpyrazone
  * Troglitazone
  * Rifapentine
  * Modafinil
  * Amiodarone
  * Anastrozole
  * Clotrimazole
  * Cyclosporine
  * Danazol
  * Delavirdine
  * Diethyldithiocarbamate
  * Diltiazem
  * Dirithromycin
  * Disulfiram
  * Entacapone (high dose)
  * Ethinyl estradiol
  * Fluoxetine
  * Fluvoxamine
  * Gestodene
  * Indinavir
  * Isoniazid
  * Metronidazole
  * Mibefradil
  * Miconazole
  * Nefazodone
  * Oxiconazole
  * Paroxetine
  * Propoxyphene
  * Roxithromycin
  * Quinidine
  * Quinine
  * Quinupristin and dalfopristin
  * Ranitidine
  * Ritonavir
  * Saquinavir
  * Sertindole
  * Sertraline
  * Troleandomycin
  * Valproic acid
  * Verapamil
  * Voriconazole
  * Zafirlukast
  * Zileuton

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2003-11; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Best objective tumor response rates (complete and partial response), based on MRIs | Up to 2 years
  Estimated ultimately as a simple binomial proportion. Estimated actuarially, using the product-limit (PL) estimate.
Time to tumor progression (TTP) | Time from study enrollment to radiographically determined tumor progression or recurrence, assessed up to 2 years
  The distribution of TTP will be analyzed using PL estimate.
Time to treatment failure (TTF) | Time from study enrollment to tumor progression, tumor recurrence, death from any cause, or occurrence of a second malignant neoplasm, assessed up to 2 years
  The distribution of TTF will be analyzed using PL estimate.
Time to death (TTD) | Time from study enrollment to death from any cause, assessed up to 2 years
  The distribution of TTD will be analyzed using PL estimate.
Incidence of adverse events graded according to NCI CTCAE version 3.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States